CLINICAL TRIAL: NCT01030094
Title: A Cross-sectional, Comparative, Multi-center Study to Investigate the Effect of Topiramate Monotherapy on Markers of Bone Mineral Metabolism and Bone Mineral Density in Premenopausal Women With Epilepsy
Brief Title: A Cross-sectional Study to Investigate the Effect of Topiramate on Bone and Mineral Metabolism in Female Participants With Epilepsy
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015856; TOP-KOR-31
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Seizures; Convulsions; Epilepsy; Osteopenia; Osteoporosis
Keywords: Topiramate; Carbamazepine; Valproic acid; Epilepsy; Bone mineral density; Monotherapy
MeSH Terms: conditions — Seizures; Epilepsy; Bone Diseases, Metabolic; Osteoporosis | interventions — Topiramate; Carbamazepine; Valproic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Topiramate: Female participants with epilepsy will be observed, who were receiving topiramate for more than one year.
  Interventions: Drug: Topiramate
- Carbamazepine: Female participants with epilepsy will be observed, who were receiving carbamazepine for more than one year.
  Interventions: Drug: Carbamazepine
- Valproic acid: Female participants with epilepsy will be observed, who were receiving valproic acid for more than one year.
  Interventions: Drug: Valproic acid
- Normal Control: Healthy female participants will be observed in Normal control group.
  Interventions: Drug: Normal control

INTERVENTIONS:
Drug: Topiramate — This is an observational study. Female participants with epilepsy will be observed, who were receiving topiramate for more than one year.
  Groups: Topiramate
Drug: Carbamazepine — This is an observational study. Female participants with epilepsy will be observed, who were receiving carbamazepine for more than one year.
  Groups: Carbamazepine
Drug: Valproic acid — This is an observational study. Female participants with epilepsy will be observed, who were receiving valproic acid for more than one year.
  Groups: Valproic acid
Drug: Normal control — This is an observational study. Healthy female participants will be observed in Normal control group.
  Groups: Normal Control

SUMMARY:
The purpose of this study is to investigate the influence of topiramate monotherapy on the bone and mineral metabolism markers, and bone density (the amount of mineral per square centimeter of bone ) in female participants with epilepsy (seizure disorder), before menopause (time in life when a woman stops having a menstrual period), as compared with healthy participants and comparative group received either carbamazepine or valproic acid monotherapy for at least last one year.

DETAILED DESCRIPTION:
This is a cross-sectional (observations or measurements made at a single point in time, usually at participant enrollment), multi-center (conducted in more than one center), and comparative study of topiramate monotherapy in female participants with epilepsy. Female participants must have received either topiramate, carbamazepine, or valproic acid monotherapy for more than one year for the treatment of epilepsy. Blood samples will be obtained from fasting participants to investigate the effect of study drug on the bone and mineral metabolism markers, and bone density compared to healthy participants and comparative group (carbamazepine and valproic acid monotherapy). Bone mineral density will be measured from the participants' lumbar spine or femur. A survey of food intake and physical activity for the participants will be performed using a standardized validated detailed questionnaire. The post-study visit (or follow up phone contact) will be performed for the occurrence of serious adverse events (SAE) for safety evaluation. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who agree to participate in this study
* Female epileptic participants
* Participants who are receiving topiramate, carbamazepine or valproic acid monotherapy for more than one year
* Participants who are using proper contraceptive method (s) or have a negative pregnancy test result

Exclusion Criteria:

* Participants with a motor function disorder
* Participants with a disease which affects their skeleton including primary hyperparathyroidism, Paget's disease, multiple myeloma, liver and kidney disorder, thyroid disease, malabsorption disorder, diabetes, and malignancies
* Participants who have taken within last one year, or are currently taking a drug which affects the bone and mineral metabolism such as vitamin D, calcium, anabolic steroids, bisphosphonates, calcitonin, glucocorticoids, and diuretics
* Voluntary or surgical postmenopausal participants
* Participants with amenorrhea for more than 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female participants with epilepsy who are receiving topiramate, carbamazepine or valproic acid monotherapy for more than one year.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Absolute Concentration of Calcium in Serum and Random Urine | 24 hours
  Bone and mineral metabolic marker represents the structure, cyclical metabolism, and hormone regulation of bone. Urinary calcium is one of the indicators of bone resorption (bone loss due to osteoclastic activity). Absolute concentration of calcium in serum and random urine will be assessed.
Absolute Concentration of 25-hydroxy Vitamin D, Osteocalcin, Carboxy-terminal Telopeptide of type 1 collagen (CTx) and Somatomedin-C (IGF-1) in Serum | 24 hours
  Osteocalcin is a vitamin K-dependent calcium-binding protein synthesized by osteoblasts and found primarily in bones. Serum osteocalcin measurements provide a noninvasive specific marker of bone metabolism. CTx is marker for bone resorption (bone loss due to osteoclastic activity). IGF-1 has growth-regulating, insulin-like, and mitogenic activities. Absolute concentration of 25-hydroxy vitamin D, osteocalcin, carboxy-terminal telopeptide of type 1 collagen (CTx) and somatomedin-C (IGF-1) in serum will be assessed.
Absolute Concentration of 1-alpha 25-dihydroxyvitamin D-3, Parathyroid Hormone (PTH) in Serum | 24 hours
  Bone and mineral metabolic marker represents the structure, cyclical metabolism, and hormone regulation of bone. 1-alpha 25-dihydroxyvitamin D-3 (vitamin D-3) and Parathyroid hormone (PTH) were assessed. The PTH maintains intracellular calcium levels in the body.
Absolute Concentration of Bone-specific Alkaline Phosphatase (BSAP) in Serum | 24 hours
  Bone and mineral metabolic marker represents the structure, cyclical metabolism, and hormone regulation of bone. Bone-specific alkaline phosphatase (BSAP) reflects formation of organic matrix in bone. Absolute concentration of BSAP in Serum will be assessed.
Absolute Concentration of Bicarbonate in Serum | 24 hours
  Bicarbonate levels in the blood are an index of the alkali reserve or buffering capacity. Difference in Bicarbonate level between topiramate, carbamazepine and valproic acid monotherapy groups will be assessed.
Absolute Concentration of Calcium in Urine in 24 Hours | 24 hours
  Absolute concentration of calcium in urine will be examined by urine test.

SECONDARY OUTCOMES:
Spine, Total hip and Femoral Neck Z-Score | 24 hours
  Z-score is number of standard deviations a participant's bone mineral density (BMD) differs from the average BMD of their age, sex, and ethnicity. Positive scores indicate BMD above the mean; Positive values are "best values" and negative values are "worst values". Z-score will be evaluated for spine, hip and femoral neck.
Percentage of Participants With Osteopenia and Osteoporosis Based on Spine T-score | 24 hours
  Osteoporosis means reduction of bone mass without alteration in the composition of bone, leading to fractures. Osteopenia is a metabolic bone disease. The T-score is a radiographic diagnosis that compares bone mineral density (BMD) to that of a "normal, healthy, 30-year-old female". The lower the T-score, the lower the BMD. A T-score of +1 to -1 is normal. A T-score decrease of -1 indicates a 10%-15% decrease in BMD. Percentage of participants with osteopenia and osteoporosis based on spine T-score will be assessed.
Percentage of Participants With Osteopenia and Osteoporosis Based on Spine Z-score | 24 hours
  Osteoporosis means reduction of bone mass without alteration in the composition of bone, leading to fractures. Osteopenia is a metabolic bone disease. The Z-score is number of standard deviations a participant's bone mineral density (BMD) differs from the average BMD of their age, sex, and ethnicity. Positive scores indicate BMD above the mean; Positive values are "best values" and negative values are "worst values". Z-score will be evaluated for spine, hip and femoral neck. Percentage of participants with osteopenia and osteoporosis based on spine Z-score will be assessed.
Absolute Concentration of Phosphorus and Creatinine in Random Urine | 24 hours
  Absolute concentration of phosphorus and creatinine in urine will be examined by urine test.
Absolute concentration of Sodium in Random Urine | 24 hours
  Absolute concentration of sodium in urine will be examined by urine test.
Absolute Concentration of Phosphorus and Creatinine in 24 Hour Urine | 24 hours
  Absolute concentration of phosphorus and creatinine in 24 hour urine will be examined by urine test.
Absolute concentration of Sodium in 24 Hour Urine | 24 hours
  Absolute concentration of sodium in 24 hour urine will be examined by urine test.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd., Korea